CLINICAL TRIAL: NCT07128524
Title: Ketone Supplementation for Opioid Craving and Withdrawal
Brief Title: Ketones for Opioid Craving
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Caron Treatment Centers (Other)
Responsible Party: Principal Investigator, Peter Manza, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00114810
Record Dates: First submitted 2025-08-13; First posted 2025-08-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; OUD; ketone; ketone supplement; ketone supplementation; craving; withdrawal
MeSH Terms: conditions — Opioid-Related Disorders; Ketosis | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Ketone Supplement (Experimental): Participants (n=25) will receive three doses of a ketone supplement drink daily for seven days.
  Interventions: Dietary Supplement: Treatment with Ketone Supplement
- Treatment with Placebo (Experimental): Participants (n=25) will receive three doses of a placebo drink daily for seven days.
  Interventions: Dietary Supplement: Treatment with Placebo

INTERVENTIONS:
Dietary Supplement: Treatment with Ketone Supplement — Participants (n=25) will receive three doses of a ketone supplement drink daily for seven days.
  Arms: Treatment with Ketone Supplement
Dietary Supplement: Treatment with Placebo — Participants (n=25) will receive three doses of a placebo drink for seven days.
  Arms: Treatment with Placebo

SUMMARY:
The goal of this clinical trial is to learn if ketone supplementation (KS) works to reduce craving for opioids for adults with opioid use disorder (OUD) undergoing in-patient acute withdrawal management. The main questions it aims to answer are:

* Does KS reduce craving for opioids in patients with opioid use disorder?
* Does KS reduce symptoms of opioid withdrawal such as low mood and pain? Researchers will compare KS to a placebo to see if KS works to reduce craving for opioids and reduce withdrawal symptoms in adults entering in-patient acute withdrawal management for opioid use disorder.

Participants will:

* Be given KS or a placebo three (3) times daily for seven (7) days
* Complete mood, pain tolerance, and subjective opioid withdrawal assessments

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Meets currents DSM-5 criteria for OUD and admitted for opioid withdrawal management treatment at Caron Treatment Center
* Willingness to provide signed, informed consent and commit to completing the procedures in the study

Exclusion Criteria:

* Current severe gastrointestinal (GI), liver, or other clinically significant physical disease that may interfere with the intake of the ketone supplement (e.g., sever inflammatory bowel disease, cirrhosis).
* Currently taking (within the past two weeks) GLP-1 receptor agonist medications, e.g. semaglutide, which can interfere with the absorption of the ketone supplement
* Currently pregnant or lactating, for people of childbearing potential
* Judged by the principal investigator. study physician, or their designee to be an unsuitable candidate for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Tonic Craving (FORCAST) total scores | Collected at baseline, and day 7
  Faceted Opioid Research Craving Assessment for Substance use Treatment (FORCAST) (Opioid Craving): A 26-item assessment of tonic craving that the person reports having felt over the prior one or two weeks. Participants indicate how much they disagree or agree with each statement on a scale that ranges from 0-6, with 0 representing "strongly disagree", 3 representing "neither agree nor disagree", and 6 representing "strongly agree". Higher scores indicate higher levels of craving. The minimum score is 0, and the maximum scores for each of the subscales are as follows: Preoccupation: 24 Negative Reinforcement: 30 Positive Reinforcement: 24 Motivation: 30 Lack of control: 24 Uneasiness: 24 Maximum total score for all subscales = 156

SECONDARY OUTCOMES:
Subjective Opioid Withdrawal | Collected at baseline and days 1-7
  Subjective Opioid Withdrawal Scale (SOWS): a 16-item patient self-report instrument to assess common subjective symptoms of craving and withdrawal. The SOWS uses a 0-4 scale for each item (0=not at all, 1=a little, 2=Moderately, 3=Quite a bit, 4=Extremely). Higher scores indicate higher levels of opioid withdrawal. Scores range from 0-64.
Pain Sensitivity (Cold Pressor Test) | collected on day 1 and day 7
  Cold Pressor Test is a well-validated measure of pain sensitivity that consistently elicits hyperalgesia in people with OUD, including those taking medications for OUD. Individuals will perform the test no later than the end of the first day of KS and again on the last day of KS. Participants plunge their dominant hand and forearm in an ice bath maintained at 5 degrees C. There are two outcomes associated with this test: pain threshold and pain tolerance. Pain threshold is the duration of time lapsed before the individual rates the sensation as painful. Pain tolerance is the duration of time the individuals keeps their arm immersed before it becomes subjectively unbearable (i.e., the individual removes their arm from the bath). Trials will be terminated if their arm is still submerged after five minutes, since pain responses on this task tend to peak by 90 seconds and diminish to below tolerance threshold within five minutes of immersion.
Desire for Drugs Questionnaire (DDQ) | collected on days 1-7
  Desires for Drugs Questionnaire (DDQ): A 14-item assessment measured on a 7-point Likert scale with 0 representing "totally disagree" and 6 representing "totally agree" and is composed of three subscales: Desire and Intention, Negative Reinforcement, and Control. A higher score indicates a higher desire for the drug.
Mood Ratings on a Visual Analogue Scale (VAS) | collected on days 1-7
  A six-item validated visual analogue scale of self-report of mood. The six items represent the three primary factors of the Profile of Mood States (happy, sad, alert, tired, relaxed, nervous) Participants will see a horizontal line with 0 on the left end and 100 on the right end and will be asked "With zero (0) meaning 'Not [Happy, Sad, etc.] At All' and 100 meaning '[Happiest/Saddest, etc.] Ever' please indicate the point on the line that represents your current state."
Chronic pain | collected at baseline and day 7
  Graded Chronic Pain Scale (GCPS-R) is a 6-item instrument that evaluates chronic pains severity (intensity and impact on life activities). Graded scores range from 0-3 (0=Chronic Pain Absent, 1=Mild Chronic Pain, 2=Bothersome Chronic Pain, 3=High Impact Chronic Pain). Higher scores indicate higher impact of chronic pain.
Mood (Positive and Negative Affect Schedule) | collected days 1-7
  Positive and Negative Affect Schedule (PANAS) is a 20 item Likert type instrument in which participants rate the extent to which they have felt specific emotions (both positive and negative) over the past week (or since they last completed the survey). The PANAS uses a 1-5 scale (1=very slightly or not at all, 2=a little, 3=moderately, 4=quite a bit, 5=extremely) for each item, with higher scores indicating a higher extent that a participant has experienced a particular emotion. Scores range from 20-100.

OTHER OUTCOMES:
Gut microbiome beta diversity | collected at baseline and day 7
  Stool samples will be collected and the beta diversity of the gut microbiome of the experimental (ketone supplement) group will be compared to the placebo group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Manza, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Caron Pennsylvania Addiction Treatment and Rehab Center, Wernersville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided